CLINICAL TRIAL: NCT04043299
Title: Birth Asphyxia in Uganda: Prevalence, Associated Factors and Effect of Intrapartum Oxygen Administration on Fetal and Early Neonatal Outcomes
Brief Title: Effect of Intrapartum Oxygen Administration on Fetal and Early Neonatal Outcomes
Acronym: Intra-O
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SHSREC 2017-051
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Fetal Distress; Birth Asphyxia
Keywords: Intrapartum oxygen administration; first stage of labour
MeSH Terms: conditions — Fetal Distress; Asphyxia Neonatorum | interventions — Oxygen; Air

STUDY DESIGN:
Intervention Model Description: The intervention group will receive 100% medical oxygen while the control group will receive medical air
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Similar gas tanks will be used for both the intervention and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive 100% oxygen at a rate of 10L/min for 15 minutes
  Interventions: Drug: 100% Oxygen
- Control (Active Comparator): This arm will receive medical air (21% oxygen) at a rate of 10 L/min for 15 minutes
  Interventions: Drug: 21% oxygen

INTERVENTIONS:
Drug: 100% Oxygen — High flow cylinder oxygen will be administered to women with fetal distress during labor
  Other Names: Medical oxygen
  Arms: Intervention
Drug: 21% oxygen — High flow cylinder packaged medical air will be administered to women with fetal distress during labr
  Other Names: Medical air
  Arms: Control

SUMMARY:
Introduction Birth asphyxia is one of leading causes of neonatal mortality in Uganda. It is associated with long term neuro-developmental complications among the babies that survive. Preventive measures for birth asphyxia intrauterine are not clearly understood and thus the need for this study.

The aim of the study is to assess the effect of intrapartum oxygen administration on fetal and early neonatal outcomes.

Methods A double-blind randomized clinical trial which will be conducted in Gulu regional referral and Kawempe National referral hospitals in Uganda. A total sample size of 1108 women in labour will be enrolled with 554 participants per group. The intervention will include administration of 10 L/min of 100% oxygen for 15 minutes to women in established labor who have signs of fetal distress with fetal heart rate of less than 120 or above 160 beats per minute. The control group will receive medical air (21% oxygen) using the same criteria. Women and babies will be followed up until 7 days after birth to document the outcomes. Statistical analysis to identify difference in outcomes between the control and intervention groups will be performed.

Ethical considerations Ethical approval and permission was received from relevant research and ethics committees. Informed consent will be sought from the participants. A data and safety monitoring board will be set up to review periodically the progress of the clinical trial study. Participants will be monitored for adverse events and severe adverse events; reporting will be done according to the research and ethics committee guidelines.

DETAILED DESCRIPTION:
Background:

Foetal distress which refers to fetal heart rate of less than 120 or more than 160 beats per minute(Pildner von Steinburg et al., 2013) during labour is one of the contributing factors to poor newborn outcomes. A proportion of these newborns will require interventions after birth such as resuscitation, oxygen therapy, antibiotics and prolonged hospital admissions. According to a retrospective study in Nigeria, 23% of foetuses diagnosed with fetal distress were born with asphyxia which is a major cause of newborn deaths(Adanikin & Awoleke, 2017). Several interventions to optimise fetal wellbeing as preparations for birth are being instituted have been suggested. These include amnio-infusion, maternal positioning, tocolysis, oxygen administration and intravenous fluid bolus(Bullens, van Runnard Heimel, van der Hout-van, & Oei, 2015; Simpson, 2007). Reviews of intrauterine resuscitation techniques have reported sufficient evidence for use of tocolysis and maternal repositioning to improve fetal pH and Apgar scores(Bullens et al., 2015; Velayudhareddy & Kirankumar, 2010). Although oxygen is used in several settings for intrauterine resuscitation(Dawood & Al-Arnous, 2002; Siriussawakul et al., 2014), its effect when used in labour for management of foetal distress remains debatable. In a Cochrane review to evaluate efficacy of oxygen administration in preventing fetal distress, only two clinical trials were found. There was evidence that the fetal arterial partial pressures of oxygen were improved by oxygen administration although there was a negative effect on pH levels. There is insufficient evidence to recommend or disprove use of oxygen for intrauterine resuscitation(Fawole & Hofmeyr, 2012). This therefore creates sufficient equipoise to undertake this study. In low resource setting where pregnant women are most likely to have anaemia, suffer from malaria and other infections, the role of oxygen for intrauterine resuscitation needs to be explored.

Aim: This study will assess the effect of administration of oxygen to women with fetal distress in the first stage of labour on fetal and early neonatal outcomes in a low resource setting.

Hypothesis: Administering 100% oxygen for 15 minutes to women with fetal distress will reduce the rate of fetal distress by 30% in the first stage of labour.

Study design: A randomised clinical trial with parallel assignment will be conducted.

Setting: The trial will take place in Gulu regional and Kawempe National referral hospitals in Uganda.

Study population: The study population will consist of pregnant women in the first stage of labour (that is between 4-10 cm cervical dilation).

Sample size: Using the Kelsey formula for sample size calculation for randomized controlled trials, with a ratio of intervention to controls of 1:1, 1108 women will be recruited.

Randomisation Block randomisation will be done to reduce the risk of bias in the study and ensure that each of the two groups has equal numbers of participant. A sequence of variable block sizes (4, 6 and 8) will be generated using STATA 15 by a statistician who will not be part of the study team.

Allocation and concealment: The allocation concealment will be done by the pharmacist in Uganda who will be in charge of storage of the control and intervention gas cylinders and dressing them with similar tamper proof jackets. The pharmacist will receive the randomization sequence from the statistician and label each masked cylinder with a set of participant serial numbers. Copies of these serial numbers will be concealed in opaque envelopes and given to research assistants.

Blinding/Masking: This will be a double blind study where the participants, the investigator, research assistants, and outcome assessors will not know the participants allocated to either intervention or control arm of the study. Unblinding of allocation will be done if the occurrence of serious adverse events increase above the study site's rates warranting investigation by the data safety monitoring board. In this case, the unblinding will be done for the data safety monitoring board (DSMB) and not to the research team.

Study procedures Women whose fetuses develop abnormal fetal heart rate on intermittent auscultation will be evaluated for presence of fetal distress by a research assistant. Diagnosis of fetal distress will be confirmed on the basis of fetal heart monitoring for 10 minutes using a Moyo fetal monitor by the trained study research assistants. A FHR below 120 or above 160 beats per minute will be considered fetal distress Standard care: All women with fetal distress will receive current standard of care which may include, encouragement for take oral fluids, administration of intravenous fluids such as Ringer's lactate, normal saline or dextrose, maternal lateral positioning and stopping the oxytocin infusion if the woman is undergoing induction or augmentation.

The intervention: Women allocated to the intervention arm will receive 100% oxygen, 10 liters per minute via non re-breather face mask for 15 minutes. The control group will receive medical air which contains 21% oxygen. 10 liters per minute via a non re-breather face mask for 15 minutes.

Monitoring and follow up: Fetal heart rate will be monitored after the intervention is commenced every 15 minutes for 1 hour or until the woman delivers the baby depending on which one comes first. After one hour of monitoring, the fetal heart rate will be monitored according to hospital protocols that is every 15 minutes if the fetal heart rate is still abnormal or every 30 minutes if it normalizes. Follow up will be done until 7 days after delivery.

Data collection Principal investigator and research assistants will collect personal, socio-demographic and pregnancy related data. Case record forms(CRFs) will be used to collect patient demographic data, maternal characteristics and results of the fetal heart rate monitoring. These forms will be filled in by the research assistants allocated to the particular shift. Data from laboratory tests will also be filled into the CRFs. A copy of results will be kept in the patient's hospital records. A study coordinator at each study site will ensure that all data for each patient has been properly captured daily and/or before the woman is discharged.

Data management Daily electronic entry will be done from the paper CRFs by the research assistants. Data will be entered into Epidata software 3.0 during the study period. This data will be checked for completeness daily and any missing data retrieved before the participants are discharged usually in 24 hours. The CRFs will be kept in a lockable cupboard placed in the labor ward with the key only accessible to the research team. The electronic data will be stored on a password protected computer accessible only by the principal investigator.

Data analysis Analysis will be according to intention to treat. Women in the control group who for one reason or another require oxygen shall not be denied the treatment but will however still be analysed according to their original assigned groups. All participants that are randomized will be analysed including those who drop out for one reason or the other. Reasons for dropout will be provided in the patient enrollment flow chart.

Data will be entered into STATA 15 software for analysis. Descriptive statistics will be computed to analyse for similarities and differences in the intervention and control group. Simple chi-squares will be used to assess differences in the study groups. The expected outcome in the two groups will be categorically analysed and proportions of participants whose fetal heart rate normalized within 30 minutes will be determined. The effect of oxygen therapy on early neonatal outcomes will also be determined using a multi-variable logistic regression model. Odds ratios will be calculated to determine associations between the outcome and predictors variables.

Quality control: Allocation concealment and blinding will be done to improve the rigor and methodological quality of the study. Fetal heart rate will be assessed objectively using the Moyo fetal heart rate monitor. Research assistants will be trained before the study commences and ongoing support supervision will be done. All procedures will follow the prescribed standard operating procedures developed in consultation will available literature. Data collected on the CRFs will be checked for completeness by the site coordinators and entered into the software regularly for cleaning. Ongoing monitoring by the study monitor and the DSMB will be done as well as visits from the ethics committee to ensure compliance with the ethical principles.

Adverse events and serious adverse events reporting Normobaric Oxygen is a category A drug for pregnant women and is therefore associated with minimal risks. Minor adverse events (AE) may include; cough, chest pain, mild dyspnea/ hypo-ventilation, malaise, nausea or tingling sensation on the skin. These signs and symptoms only occur if the oxygen is administered for more than 6 hours.

Serious adverse events (SAE) will include but not limited to, serious maternal complications such as antepartum hemorrhage, postpartum hemorrhage, disseminated intravascular coagulopathy (DIC), still birth, neonatal death, and maternal death. The principal investigator(PI) will be notified of any AE and SAE within 48 hours. In case of a SAE, it will be reported by the PI to the primary ethics committee within 7 days. According to the Uganda National council of science and technology guidelines, SAEs will be reported to the DSMB, National drug authority and the ethics committee.

Ethical considerations Ethical approval was obtained from the higher degrees research and ethics (HDREC) committee at the School of Health Sciences, Makerere University and the National Council for higher education. Approval was also received from the Uganda National drug authority and administrative clearances from both study sites. Verbal and written informed consent will be obtained from participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women in active first stage of labor who develop fetal distress will be included

Exclusion Criteria:

* Women in labor with critical conditions such as eclampsia, chronic heart disease, chronic lung disease and chronic renal failure
* Women in preterm labor
* Those taking Bleomycin and Amiodarone medications

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1108 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Normalization of the fetal heart rate | 30 minutes
  The fetal heart rate will be between 120 to 160 beats per minute

SECONDARY OUTCOMES:
Birth Asphyxia | At 5 minutes after birth
  Five minute Apgar score of less than 7 at 5 minutes. Apgar Score refers to Appearance, pulse, grimace, activity and respiration. Each of these 5 elements are scored from 0-2 where by 0 is the worst score meaning absence of the parameter while 2 is the best score. A total of 0 means that the newborn has no signs of life, 1-6 refers to an infant with asphyxia while infants with scores of 7 to 10 are considered normal.
Hypoxic Ischemic encephalopathy | 24 hours and 7 days after birth
  Hypoxic ischemic encephalopathy defined by Thompson Scores of 15 or more. This score is made of 9 signs assessed on a scale of 0-3. These are tone, level of consciousness, fits, posture, moro reflex, grasp reflex, suck, respiration and fontanel. Tone, level of consiciousness and posture are scored on a scale of 0-3 while the rest are scored on a scale of 0-2. A score of 0 for each individual item means normal while 2 or 3 refers to more severe problems. The lower the score, the better for a newborn.The maximum total score is 22 and scores of less than 10 are considered normal. However in this study, we shall consider scores of 15 or more as hypoxic ischemic encephalopathy.
Neonatal Acidosis | Within 5 minutes of birth
  Neonatal acidosis defined by cord artery lactate of more than 5.5mmol/l taken after delivery
Status of newborn | 7 days after birth
  Status of newborn indicating whether baby is alive or dead

CONTACTS AND LOCATIONS:
Overall Officials: James K Tumwine, PhD, Study Director — Makerere University
Locations (1):
- Kawempe National Referral Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared with other researchers on request.

REFERENCES:
- [Background] Garite TJ, Simpson KR. Intrauterine resuscitation during labor. Clin Obstet Gynecol. 2011 Mar;54(1):28-39. doi: 10.1097/GRF.0b013e31820a062b. PMID 21278499
- [Background] Simpson KR. Intrauterine resuscitation during labor: review of current methods and supportive evidence. J Midwifery Womens Health. 2007 May-Jun;52(3):229-37. doi: 10.1016/j.jmwh.2006.12.010. PMID 17467589
- [Background] Bullens LM, Moors S, van Runnard Heimel PJ, van der Hout-van der Jagt MB, Oei SG. Practice variation in the management of intrapartum fetal distress in The Netherlands and the Western world. Eur J Obstet Gynecol Reprod Biol. 2016 Oct;205:48-53. doi: 10.1016/j.ejogrb.2016.08.012. Epub 2016 Aug 16. PMID 27566222
- [Background] Adanikin AI, Awoleke JO. Clinical suspicion, management and outcome of intrapartum foetal distress in a public hospital with limited advanced foetal surveillance. J Matern Fetal Neonatal Med. 2017 Feb;30(4):424-429. doi: 10.1080/14767058.2016.1174991. Epub 2016 Apr 25. PMID 27050656
- [Background] Fawole B, Hofmeyr GJ. Maternal oxygen administration for fetal distress. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD000136. doi: 10.1002/14651858.CD000136.pub2. PMID 23235574
- [Background] Weeke LC, Vilan A, Toet MC, van Haastert IC, de Vries LS, Groenendaal F. A Comparison of the Thompson Encephalopathy Score and Amplitude-Integrated Electroencephalography in Infants with Perinatal Asphyxia and Therapeutic Hypothermia. Neonatology. 2017;112(1):24-29. doi: 10.1159/000455819. Epub 2017 Feb 17. PMID 28208138
- [Background] Vernon G, Alfirevic Z, Weeks A. Issues of informed consent for intrapartum trials: a suggested consent pathway from the experience of the Release trial [ISRCTN13204258]. Trials. 2006 May 11;7:13. doi: 10.1186/1745-6215-7-13. PMID 16689989
- [Background] Lawton J, Snowdon C, Morrow S, Norman JE, Denison FC, Hallowell N. Recruiting and consenting into a peripartum trial in an emergency setting: a qualitative study of the experiences and views of women and healthcare professionals. Trials. 2016 Apr 11;17:195. doi: 10.1186/s13063-016-1323-3. PMID 27066777
- [Background] Pildner von Steinburg S, Boulesteix AL, Lederer C, Grunow S, Schiermeier S, Hatzmann W, Schneider KT, Daumer M. What is the "normal" fetal heart rate? PeerJ. 2013 Jun 4;1:e82. doi: 10.7717/peerj.82. Print 2013. PMID 23761161
- [Background] Siriussawakul A, Triyasunant N, Nimmannit A, Ngerncham S, Hirunkanokpan P, Luang-Aram S, Pechpaisit N, Wangdee A, Ruangvutilert P. Effects of supplemental oxygen on maternal and neonatal oxygenation in elective cesarean section under spinal anesthesia: a randomized controlled trial. Biomed Res Int. 2014;2014:627028. doi: 10.1155/2014/627028. Epub 2014 Feb 20. PMID 24696860
- [Background] Thorp JA, Trobough T, Evans R, Hedrick J, Yeast JD. The effect of maternal oxygen administration during the second stage of labor on umbilical cord blood gas values: a randomized controlled prospective trial. Am J Obstet Gynecol. 1995 Feb;172(2 Pt 1):465-74. doi: 10.1016/0002-9378(95)90558-8. PMID 7856671
- [Background] Dawood MA, Al-Arnous MA. The Effect of Maternal Oxygen Adminstration During The Second Stage of Normal Vaginal Delivery Or During Cesarean Section Under General Anaesthesia On Umblical Cord Blood Gases and Acid-Base State. Alexandria Journal of Pediatrics. 2002;16(2):233.
- [Background] Casey BM, McIntire DD, Leveno KJ. The continuing value of the Apgar score for the assessment of newborn infants. N Engl J Med. 2001 Feb 15;344(7):467-71. doi: 10.1056/NEJM200102153440701. PMID 11172187
- [Background] Morales P, Bustamante D, Espina-Marchant P, Neira-Pena T, Gutierrez-Hernandez MA, Allende-Castro C, Rojas-Mancilla E. Pathophysiology of perinatal asphyxia: can we predict and improve individual outcomes? EPMA J. 2011 Jun;2(2):211-30. doi: 10.1007/s13167-011-0100-3. Epub 2011 Jul 26. PMID 23199150